CLINICAL TRIAL: NCT05729009
Title: The Evolution of Systemic Microvascular Reactivity in Heart Transplant Patients
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Principal Investigator, National Institute of Cardiology, Laranjeiras, Brazil
Other Study IDs: 45581521.0.0000.5272
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- heart transplantation
  Interventions: Diagnostic Test: skin microvascular reactivity

INTERVENTIONS:
Diagnostic Test: skin microvascular reactivity — Laser-based method for evaluating non-invasive, operator-independent systemic microvascular function that detects microvascular flow in the skin for the evaluation of systemic vascular endothelial function.

SUMMARY:
The evolution of systemic microvascular reactivity may aid in the comprehension of cardiovascular physiology in heart transplantation patients, and possibly suggest the non-invasive evaluation of skin microcirculation as an ancillary tool in the clinical evaluation of these patients.

DETAILED DESCRIPTION:
Introduction: Systemic microvascular reactivity (MR) is an essential component of cardiovascular physiology, being studied through non-invasive techniques in readily accessible body regions, such as the skin surface. Heart transplant (HT) is a treatment considered to selected patients, with advanced heart failure. The main cause of long-term mortality after HT is graft vascular disease (GVD), a condition which starts with endothelial dysfunction. To know the evolution of systemic MR in patients subjected to HT can help to find prognostic factors. Objective: The present study aims to perform the prospective evaluation of systemic MR in adult patients, before and two years after HT, at a quaternary hospital, correlating the findings with clinical variables. Methods: Systemic MR will be evaluated in the skin of the forearm using laser speckle contrast imaging with acetylcholine (ACh) iontophoresis, followed by postocclusive reactive hyperemia (PORH), before and after HT. Measurements will be correlated to patient clinical profile, hemodynamic and echocardiographic data. Expected results: The evolution of systemic MR may aid in the comprehension of cardiovascular physiology in HT patients, and possibly suggest the non-invasive evaluation of skin microcirculation as an ancillary tool in the clinical evaluation of these patients.

ELIGIBILITY:
Inclusion Criteria:

* capability to understand the objectives of the research and to fulfill the Term of Consent

Exclusion Criteria:

* Pregnancy, acute infection diagnosis, use of circulatory assistance devices

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult individuals from the cohort of heart failure patients under evaluation for heart transplantation, at the National Institute of Cardiology, Rio de Janeiro, Brazil
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Baseline and post-iontophoresis of acetylcholine endothelium-dependent skin microvascular reactivity | Microvascular reactivity will be evaluated 20-minute rest in the supine position in a temperature-controlled room.
  Evaluation of systemic microvascular reactivity induced by endothelium-dependent agents. Microvascular reactivity will be evaluated using a non-invasive and operator -independent methodology, named laser speckle contrast imaging, coupled with skin iontophoresis of vasodilator agents. Cutaneous microvascular flow will be measured in arbitrary perfusion units, divided by mean arterial pressure, to yield cutaneous vascular conductance.

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo Tibiriçá, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No